CLINICAL TRIAL: NCT03000790
Title: Clinical Evaluation of Lingual Ring Splint For Management Anterior Disc Displacement With Reduction (Pilot Study Clinical Trial)
Brief Title: Evaluation Lingual Ring Splint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Nassar, Dentist at ministry of health, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CairoLRS
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: TMJ Disc Disorder
Keywords: Anterior disc displacement; TMD therapy; internal derangement; Lingual Ring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lingual Ring Splint (Experimental): A polyvinyl (polypropylene) material was chosen, which is biocompatible, nontoxic, hypoallergenic, and has a hardness of about 60-70 Shore, The thickness of 3 mm in the occlusive active portion and 2 mm in the other parts was constructed.
  The lingual ring consists of Two lateral genal shields that are vertical and symmetric, and have a right- and left-of-oval form, Two interocclusive levels with a roughly triangular form, but with round angles also right and left symmetric, double arch superior arch and inferior arch will make the Ring around the tongue
  Interventions: Device: Lingual Ring Splint

INTERVENTIONS:
Device: Lingual Ring Splint — A polyvinyl (polypropylene) material was chosen, which is biocompatible, nontoxic, hypoallergenic, and has a hardness of about 60-70 Shore, The thickness of 3 mm in the occlusive active portion and 2 mm in the other parts was constructed.
  The lingual ring consists of Two lateral genal shields that are vertical and symmetric, and have a right- and left-of-oval form, Two interocclusive levels with a roughly triangular form, but with round angles also right and left symmetric, double arch superior arch and inferior archwill make the Ring around the tongue

SUMMARY:
To evaluate the effectiveness of Lingual Ring Splint For Management of Anterior Disc Displacement With Reduction

DETAILED DESCRIPTION:
To evaluate the effectiveness of Lingual Ring Splint For Management of Anterior Disc Displacement With Reduction.

PICO P- Patient with symptomatic anterior disc displacement with reduction . I- use of Michigan splint C- use of anterior repositioning splint (ARS) . O- Clinical outcome. Pain relief and improvement of mouth opening , lateral excursion and protrusion

Outcome:

* 1ry outcome: Patients' subjective pain experience. Each patient will be asked to rate his or her current and worst pain intensity on numerical rating scale (NRS) of 0-10 with zero being no pain and ten corresponds to the worst pain that the patient ever had.
* 2ry outcome:

  1. Maximum mouth opening (MMO). Assessment of MMO will be performed by measuring the distance in mm between the incisal edges of the upper and lower central incisors using a ruler.
  2. lateral excursion . Assessment of lateral excursion will be performed by measuring the distance in mm between midline of upper and lower jaws
  3. protrusion. The distance in mm from the incisal edge of the maxillary central incisor to the incisor edge of the mandibular incisor will measured in the maximum protruded position.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient from 15 to 50 years old.
* Report of pain in preauricular region, in the last 30 days, worsened by functional activities, such as chewing and talking.
* Presence of disc displacement with reduction, arthralgia and joint clicking that occurred at both middle to late opening and late closing (near maximum cuspation) and pain in the TMJ area aggravated by jaw movement and function.
* positive diagnosis of unilateral or bilateral anterior disc displacement with reduction by means of magnetic resonance imaging (MRI).

Exclusion Criteria:

* Individuals with a recent history of trauma in the face and/or neck area.
* Individuals with systemic diseases that can affect TMJ.
* History of TMJ surgery.
* Individuals with dental pain.
* Individuals with myofascial pain, disc displacement with reduction or osteoarthritis.
* Individuals under dental or TMD management.
* Individuals wearing full or partial dentures.
* Individuals with major psychological disorders.
* Nonreducing dislocations of the articular disk in the acute form of TMD
* Consequences of condoyle fractures and/or fracture of another maxillofacial zone.
* In therapy for the same pathologies.
* Articular pathologies of systemic nature (e.g., rheumatoid arthritis, arthrosis, psoriasis arthritis).
* Well-known pathologies of neurologic and/or psychic nature and other forms of migraine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Patients' subjective pain experience. | 3 months
  Each patient will be asked to rate his or her current and worst pain intensity on numerical rating scale (NRS) of 0-10 with zero being no pain and ten corresponds to the worst pain that the patient ever had.

SECONDARY OUTCOMES:
Maximum mouth opening. | 3 months
  measuring the distance between the incisal edges of the upper and lower central incisors using a ruler.Unit:mm
Lateral excursion. | 3 months
  measuring the distance between midline of upper and lower jaws . Unit: mm
Protrusion. | 3 months
  The distance in mm from the incisal edge of the maxillary central incisor to the incisor edge of the mandibular incisor will measured in the maximum protruded position.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Galal, MD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srivastava R, Jyoti B, Devi P. Oral splint for temporomandibular joint disorders with revolutionary fluid system. Dent Res J (Isfahan). 2013 May;10(3):307-13. PMID 24019797
- [Background] Seifeldin SA, Elhayes KA. Soft versus hard occlusal splint therapy in the management of temporomandibular disorders (TMDs). Saudi Dent J. 2015 Oct;27(4):208-14. doi: 10.1016/j.sdentj.2014.12.004. Epub 2015 Jun 25. PMID 26644756
- [Background] Conti PC, Correa AS, Lauris JR, Stuginski-Barbosa J. Management of painful temporomandibular joint clicking with different intraoral devices and counseling: a controlled study. J Appl Oral Sci. 2015 Oct;23(5):529-35. doi: 10.1590/1678-775720140438. Epub 2015 Jul 21. PMID 26200526
- [Background] Lee HS, Baek HS, Song DS, Kim HC, Kim HG, Kim BJ, Kim MS, Shin SH, Jung SH, Kim CH. Effect of simultaneous therapy of arthrocentesis and occlusal splints on temporomandibular disorders: anterior disc displacement without reduction. J Korean Assoc Oral Maxillofac Surg. 2013 Feb;39(1):14-20. doi: 10.5125/jkaoms.2013.39.1.14. Epub 2013 Feb 21. PMID 24471012
- [Background] Liu J, Mu H, Wang Z, Lan J, Zhang S, Long X, Zhang D. Joint cavity injection combined with manual reduction and stabilization splint treatment of anterior disc displacement. Int J Clin Exp Med. 2015 Apr 15;8(4):5943-8. eCollection 2015. PMID 26131189
- [Background] Muhtarogullari M, Avci M, Yuzugullu B. Efficiency of pivot splints as jaw exercise apparatus in combination with stabilization splints in anterior disc displacement without reduction: a retrospective study. Head Face Med. 2014 Oct 9;10:42. doi: 10.1186/1746-160X-10-42. PMID 25300939
- [Background] Rampello A, Falisi G, Panti F, DI Paolo C. A new aid in TMD Therapy: the Universal Neuromuscular Immediate Relaxing appliance "UNIRA". Oral Implantol (Rome). 2010 Jan;3(1):20-32. Epub 2010 Nov 19. PMID 23285377